## Data analysis

In the evaluation of the data, in addition to descriptive statistical methods (e.g., percentage, frequency, mean, and standard deviation), the chi-square test and Student's t-test were used in the comparison of the qualitative data. The results were evaluated at a significance level of p <0.05.

The dependent variables of the study are the pain score averages of the pregnant women, the duration of the latent, active and transition phases of labour, and the anxiety level score. The independent variables of the study are the pregnant women's age, educational status, working status, and prenatal educational status, as well as the educational status of the husbands of the pregnant women, their willingness to become pregnant and the willingness to serve as controls before labour.